CLINICAL TRIAL: NCT06466226
Title: Incidence of Complications Associated With Multiple Central Venous Accesses in the Internal Jugular Vein: a Randomized Multicenter Non-inferiority Clinical Trial
Brief Title: Complications Associated With Multiple Central Venous Accesses in the Internal Jugular Vein
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 75871523.2.0000.5530
Record Dates: First submitted 2024-05-17; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Central Venous Catheters; Catheter Complications; Catheter Related Complication
Keywords: central venous access; complications; major surgery

STUDY DESIGN:
Masking Description: No masking is possible considering the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Multiple central venous lines in two sites separately
  Interventions: Procedure: Multiple central venous lines in two sites separately
- Group 2 (Experimental): Multiple central venous lines in a single internal jugular vein
  Interventions: Procedure: Multiple central venous lines in one site (internal jugular vein)

INTERVENTIONS:
Procedure: Multiple central venous lines in two sites separately — Patients with two central venous lines in two sites separately (two central venous sites).
  Arms: Group 1
Procedure: Multiple central venous lines in one site (internal jugular vein) — Patients with two concomitant central venous lines in a single internal jugular vein (one central venous site).
  Arms: Group 2

SUMMARY:
Patients at risk of significant intraoperative blood loss and/or potential hemodynamic instability often necessitate the placement of two or more central venous catheters, including large bore catheters. In tertiary hospitals, anesthesiologists frequently encounter patients undergoing major surgeries such as liver transplantation, lung transplantation, cardiac surgery, and vascular surgery, who require multiple central venous punctures as part of routine anesthetic management. However, most review and consensus articles do not directly address the utilization of multiple catheters in the same venous site, nor establish formal recommendations regarding this practice. The latest consensus on central venous access from the American Association of Anesthesiologists (ASA), published in 2012, briefly touches upon some aspects related to this practice but does not outline any contraindications. Thus, the investigators have identified a gap in evidence and robust prospective studies addressing the use of more than one catheter in the same site for central venous access. This lacuna underscores the importance of conducting a controlled clinical study in our institutions to establish the efficacy and safety of this approach in the perioperative context. The present study aims to evaluate the incidence of mechanical complications (such as dysrhythmias, arterial puncture, hematoma, pneumothorax/hemothorax, insertion failure, or inadequate positioning) within the first 24 hours after double puncture of the internal jugular vein compared to puncture of two distinct central vessels, in patients undergoing multiple central venous accesses during major surgeries. This study will be designed as a prospective, randomized, non-inferiority, open, parallel clinical trial with two groups for patient allocation. Patients identified for multiple central venous accesses as part of preoperative anesthetic planning will be randomly allocated to either receive two central venous accesses in two separate sites (Group I or control group) or two concurrent central venous accesses in a single internal jugular vein (Group II or intervention group). Only adult patients classified as ASA I to IV (over 18 years old), scheduled for major surgery, will be eligible for inclusion.

DETAILED DESCRIPTION:
Patients at risk of significant intraoperative blood loss and/or potential hemodynamic instability often necessitate the placement of two or more central venous catheters, including large bore catheters. In tertiary hospitals, we frequently encounter patients undergoing major surgeries such as liver transplantation, lung transplantation, cardiac surgery, and vascular surgery, who require multiple central venous punctures as part of routine anesthetic management. However, most review and consensus articles do not directly address the utilization of multiple catheters in the same venous site, nor do they establish formal recommendations regarding this practice. The latest consensus on central venous access from the American Association of Anesthesiologists (ASA), published in 2012, briefly touches upon some aspects related to this practice but does not outline any contraindications. This consensus primarily references the only comparative and prospective study conducted by Reeves and colleagues in 1995, which compared the passage of multiple central venous catheters in a single site (right internal jugular vein) with placements in different sites.

Thus, the investigators have identified a gap in evidence and robust prospective studies addressing the use of more than one catheter in the same site for central venous access. This lacuna underscores the importance of conducting a controlled clinical study in our institutions to establish the efficacy and safety of this approach in the perioperative context.

Our study aims to evaluate the incidence of mechanical complications (such as dysrhythmias, arterial puncture, hematoma, pneumothorax/hemothorax, insertion failure, or inadequate positioning) within the first 24 hours after double puncture of the internal jugular vein compared to puncture of two distinct central vessels, in patients undergoing multiple central venous accesses during major surgeries.

The study will be designed as a prospective, randomized, non-inferiority, open, parallel clinical trial with two groups for patient allocation. Patients identified for multiple central venous accesses as part of preoperative anesthetic planning will be randomly allocated to either receive two central venous accesses in two separate sites (Group I or control group) or two concurrent central venous accesses in a single internal jugular vein (Group II or intervention group). The preferred site for the second central venous access in Group I will be the subclavian vein.

Only adult patients classified as ASA I to IV (over 18 years old), scheduled for major surgery, will be eligible for inclusion. Surgical procedures considered for patient allocation include cardiac surgeries, vascular surgeries, major abdominal or thoracic surgeries, liver transplants, and lung transplants. Inclusion criteria specify patients with anesthetic planning for the insertion of at least two central venous catheters.

The primary hypothesis of this study is that the incidence of mechanical complications (cardiac arrhythmias, arterial puncture, hematoma, pneumothorax/hemothorax, catheter insertion failure or inadequate catheter positioning) is equivalent with two punctures in the internal jugular vein when compared to punctures in two different central vessels (internal jugular vein and subclavian and/or femoral vein).

The secondary hypotheses of this study are that the incidence of catheter-related infection, catheter malfunction, and puncture site thrombosis is lower with two punctures in the internal jugular vein when compared to punctures in two different central vessels (internal jugular vein and subclavian and/or femoral).

The study will be designed as a prospective, randomized, non-inferiority, open, parallel clinical trial with two groups for patient allocation. Patients who, according to preoperative anesthetic planning, have indications for multiple central venous accesses (i.e., patients with indications for 2 concomitant central venous catheters) will be randomly allocated to two central venous accesses in two sites separately ( Group I or control group) or two concomitant central venous accesses in a single internal jugular vein (Group II or intervention group). The preferred site for the second group I central venous access is the subclavian.

In this study, adult patients scheduled to undergo major surgery at the Hospital de Clínicas de Porto Alegre, Santa Casa de Porto Alegre and Hospital Nossa Senhora da Conceição will be included. All hospitals involved will have equivalent importance, varying participation according to the number of surgeries performed in the institutions.

Only adult ASA I to IV patients (over 18 years old), scheduled to undergo major surgery in the aforementioned hospitals, will be included.

The surgical procedures considered in this study for patient allocation include: cardiac surgeries, vascular surgeries, major abdominal or thoracic surgeries, liver transplants and lung transplants. Only patients with anesthetic planning for insertion of at least two central venous catheters will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preanesthetic planning for insertion of at least two central venous catheters.
* Adult ASA I to IV patients (over 18 years old), scheduled to undergo cardiac surgeries, vascular surgeries, major abdominal or thoracic surgeries, liver transplants and lung transplants.

Exclusion Criteria:

* Patients with a previous history of central venous thrombosis or central venous stenosis will be excluded from the research protocol.
* Patients without preanesthetic planning insertion of at least two central venous catheters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite mechanical complications | Intraoperative
  The main outcome is to evaluate the incidence of mechanical complications (dysrhythmias, arterial puncture, hematoma, pneumothorax/hemothorax, insertion failure or inadequate positioning) in the first 24 hours after double puncture of the internal jugular vein compared to puncture of two distinct central vessels, in patients undergoing more than one central venous access in major surgeries.

SECONDARY OUTCOMES:
Incidence of catheter-related infection | Up to 30 days after surgery
  To evaluate the incidence of catheter-related infection (central line-associated bloodstream infections - CLABSI) after double puncture of the internal jugular vein compared to puncture of two distinct central vessels, in patients undergoing more than one central venous access in surgery. large.
Incidence of central venous catheter malfunction | Up to 30 days after surgery
  To evaluate the incidence of central venous catheter malfunction after double puncture of the internal jugular vein compared to the puncture of two different central vessels, in patients undergoing more than one central venous access in major surgeries.
Insertion time of a central venous catheter | Intraoperative (during central venous line insertion)
  To evaluate the insertion time of a central venous catheter after double puncture of the internal jugular vein compared to the puncture of two different central vessels, in patients undergoing more than one central venous access in major surgeries.
Number of attempts to pass each catheter | Intraoperative (during central venous line insertion)
  To evaluate the number of attempts to pass each catheter after double puncture of the internal jugular vein compared to the puncture of two different central vessels, in patients undergoing more than one central venous access in major surgeries.
Incidence of venous thrombosis within 30 days | Up to 30 days after surgery
  To evaluate the incidence of venous thrombosis within 30 days related to double puncture of the internal jugular vein compared to puncture of two different central vessels, in patients undergoing more than one central venous access in major surgeries.

CONTACTS AND LOCATIONS:
Overall Officials: Andre P Schmidt, MD, Principal Investigator — Hospital Nossa Senhora da Conceição

IPD SHARING:
Plan to Share IPD: No